CLINICAL TRIAL: NCT06312527
Title: Efficacy of a Soft Silicone Dressing to Prevent Scarring After Bilateral Total Knee Arthroplasty: A Randomized Paired Controlled Trial.
Brief Title: Mepiform in Simultaneous Bilateral TKA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University Hospital (Other)
Responsible Party: Principal Investigator, Yot Tanariyakul, Dr., Thammasat University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TUH Mepiform TKA
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Scar Prevention
Keywords: Scar prevention; total knee arthroplasty; Silicone dressing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Silicone dressing (Experimental): Apply silicone dressing after wound completely healed. Changing the dressing sheet every 7 days by Close the silicone cover for 10 weeks.
  Interventions: Device: Silicone dressing
- No intervention (No Intervention): Do not apply silicone dressing

INTERVENTIONS:
Device: Silicone dressing — Participant will apply silicone dressing at 2 weeks after TKA on one side of knee.
  Silicone dressing will change every week until 12 week postoperative.
  Arms: Silicone dressing

SUMMARY:
The goal of this RCT is comparing efficacy of silicone dressing in scar preventing after simultaneous bilateral total knee arthroplasty.

The main question[s] it aims to answer are:

* Does silicone dressing can prevent scar formation after total knee arthroplasty?
* Does silicone dressing have similar functional outcomes and complications after total knee arthroplasty? Participants will apply silicone dressing after wound healed and apply for 10 weeks. Researchers will compare to the other side that is no intervention.

DETAILED DESCRIPTION:
1. After the patient has passed the above selection criteria A team of non-surgery investigators will now describe the program in detail, the benefits and risks of the program. If the patient voluntarily agrees to participate in the program. The patient will sign the statement in writing and they can ask questions. The patients had to pass the selection criteria and be excluded from the research.
2. Record personal information about the patient's surgery, including age, sex, weight, height, knee deformities and knee severity before surgery. History of scar formation on the body (hypertrophic scar or keloid)
3. The range of motion of the knee before surgery was assessed by physical examination by using the Goniometer by the research assistant and assessing the knee functional ability score. Using the Forgotten joint score and Modified WOMAC score assessment form.
4. Joint replacement surgery for both knees using the same type of prosthetic knee. After the surgery, the wound was sutured by a joint reconstructive fellowship by sewing all 3 layers consisting of the first layer is sutured with vicryl 1/0 threads, with the upper half of the knee above the center of the patella sutured (interrupt suture), and the lower half sutured continuously (continuous locking suture). The second layer is sutured under the skin(subcutaneous suture) by stitching. The tissues are brought close together using Vicryl 1/0 threads and continuous concealed cosmetic suture using 3rd layer of Vicryl 2/0 threads. Skin closure using Monosyn 4/0 threads and covered with Leukostrip sticky tape, after which the wound was covered with an Opsite Dressing. All patient will be recommend the same standard care after discharge. Wound will be cover the with an Opsite dressing and if there leakage or water into the wound. A dry dressing is recommended, followed by an Opsite dressing.
5. Take care after surgery by giving pain medication. The standard postoperative physical therapy was the same in all patients
6. Follow-up at approximately 2 weeks after surgery. After the wound has been opened and the tape has been removed. The surgeon evaluates the wound after surgery. If there are no complications of the surgical wound. The envelope will be opened according to the researcher's number. which is randomly generated using a computer to see which side will receive a silicone sheet dressing (soft-silicone dressing, Mepiform®, Mölnlycke Health Care AB, Gothenburg, Sweden), which side does not require closure. To care for the wound after 2 weeks, the wound can be cleaned with water or soap like normal skin on both sides.
7. The patient was allowed range of motion exercise and knee motion were recorded.
8. The patient will be taught how to use the silicone sheet. By covering the entire surgical wound at least 1 cm and closing it in the knee bend approximately 30 degrees, the wound must be closed 24 hours a day by taking it out when taking a shower 1-2 times a day, changing the dressing sheet every 7 days by Close the silicone cover for 10 weeks. As a study by Thomas A, et al9 recommends covering the wound dressing to prevent postoperative scarring. At least for a period of 2 months, errors will be controlled with a silicone sheet closure instruction sheet for all patients. including identifying the side that covers the silicone sheet.
9. Appointment for follow-up treatment of patients after surgery Follow-up assessments will be made at approximately 6 weeks, 3 months, 6 months and 1 year after surgery. The research assistant measured the flexion range of the knee joint and assessing the function of the knee joint. The scar will be assessed by a dermatologist which will not know which side will be the side that has been using the silicone cover throughout the evaluation. Including the evaluation of wound complications such as split wounds, thrombosis around the surgical wound, Abscesses due to stitch abscess and other complications such as Deep vein thrombosis. If such complications, Research participants will be excluded from the study and will receive standard treatment by the research physicians team.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 50-80 years
2. The participant who undergo simultaneous bilateral total knee arthroplasty.
3. The participant can understand and give consent to participate in the project.

Exclusion Criteria:

1. The participants had previous knee surgery
2. The participants have had a scar on the knee before getting the surgery. 3. Periprosthetic joint infection.

4. There are other complications of the surgical wound, such as split wound, thrombosis around the surgical wound. Abscess caused by stitches (stitch abscess) 5. Deep vein thrombosis (DVT)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Vancouver Scar Scale | 6week, 3month, 6month, 1 year
  Vancouver Scar Scale evaluate by dermatologist (point) Range from 0-13 (0 mean best, 13 mean worst)

SECONDARY OUTCOMES:
Range of motion | 6week, 3month, 6month, 1 year
  evaluate by long arm goniometer (degree)
Forgotten joint score | 6week, 3month, 6month, 1year
  Forgotten joint score (point) (range 0-100, 0 mean worst, 100 mean best)
modified WOMAC score | 6week, 3month, 6month, 1year
  modified WOMAC score (point) (range 0-96, 0 mean best, 96 mean worst)
Scar pain | 6week, 3month, 6month, 1year
  evaluate by visual analog scale (point) (0-10, 0 mean best, 10 mean worst)
Scar itching | 6week, 3month, 6month, 1year
  evaluate by visual analog scale (point) (0-10, 0 mean best, 10 mean worst)
Complications | 6week, 3month, 6month, 1year
  Wound complication ex deep joint infection, surgical site infection, wound dehiscence

CONTACTS AND LOCATIONS:
Overall Officials: Yot Tanariyakul, M.D., Principal Investigator — Department of orthopedics
Locations (1):
- Thammasat University, Khlong Luang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kong CG, Kim GH, Kim DW, In Y. The effect of topical scar treatment on postoperative scar pain and pruritus after total knee arthroplasty. Arch Orthop Trauma Surg. 2014 Apr;134(4):555-9. doi: 10.1007/s00402-014-1942-7. Epub 2014 Feb 9. PMID 24509938